CLINICAL TRIAL: NCT06391151
Title: Effect of Obstructive Sleep Apnea (OSA) Resulting From Chronic Tonsillitis on Pregnancy Outcomes
Brief Title: Effect of OSA Resulting From Chronic Tonsillitis on Pregnancy Outcomes
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Xiaowan Du, Principal Investigator, Peking University First Hospital
Other Study IDs: PKUFH ENT TLP V1.0
Record Dates: First submitted 2024-04-24; First posted 2024-04-30 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Obstructive Sleep Apnea; Chronic Tonsillitis; Pregnancy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: exposure: OSA resulting from chronic tonsillitis — exposure: OSA resulting from chronic tonsillitis

SUMMARY:
This cohort study aims to investigate the impact of obstructive sleep apnea hypopnea syndrome (OSA) resulting from chronic tonsillitis on pregnancy outcomes. The hypothesis posits that chronic tonsillitis-induced OSA may exacerbate pregnancy complications and increase the risk of adverse pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women confirmed with chronic tonsillitis by clinical diagnosis and presenting symptoms.
* Pregnant women with a confirmed diagnosis of OSA based on polysomnography or other validated sleep monitoring techniques.
* Pregnant women who are willing to participate in the study and provide informed consent.

Exclusion Criteria:

* Pregnant women with other respiratory or sleep disorders that may confound the diagnosis of OSA.
* Pregnant women with severe comorbidities or medical conditions that may significantly impact pregnancy outcomes.
* Pregnant women who have undergone surgical treatment for chronic tonsillitis or OSA during the study period.
* Pregnant women who refuse to participate in the study or are unable to provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnancy
Study Population: Pregnant women who have established prenatal care records and undergone antenatal check-ups at PKUFH
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
preterm birth rate | 10 months

SECONDARY OUTCOMES:
delivery methods | 10 months

OTHER OUTCOMES:
pregnancy complications | 10 months
neonatal birth weight | 10 months
  birth weight of newborns measured in grams
neonatal length | 10 months
  length of newborns measured in centimeters
Apgar score of newborns | 10 months
  The Apgar score consists of five main indicators: skin color, heart rate, response to stimulation, muscle tone, and respiration. Each indicator is scored from 0 to 2, with a total score of 10. This scoring method serves as a guiding tool for the resuscitation of newborns with asphyxia and could provide a degree of predictive value for the neurological development of infants in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaowan Du, Study Director — Peking University First Hospital

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be provided upon request.